CLINICAL TRIAL: NCT06233617
Title: Dexamethasone vs. Dexmedetomidine for ESPB in Pain Management After Spine Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3/2024
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Spinal Fusion; Spine Disease; Spinal Stenosis; Erector Spinae Plane Block
MeSH Terms: conditions — Spinal Diseases; Spinal Stenosis | interventions — Sodium Chloride; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator): 0.2% ropivacaine for erector spinae plane block
  Interventions: Drug: 0.9% Sodium Chloride Injection
- Dexamethasone (Active Comparator): 0.2% ropivacaine + 4mg Dexamethasone for erector spinae plane block
  Interventions: Drug: Dexamethasone 4 Mg/mL Injectable Solution
- Dexmedetomidine (Active Comparator): 0.2% ropivacaine + 50ug Dexmedetomidine for erector spinae plane block
  Interventions: Drug: Dexmedetomidine injection

INTERVENTIONS:
Drug: 0.9% Sodium Chloride Injection — biliteral administration of 20ml of 0,2% ropivacaine + 2ml 0.9% sodium chloride for the erector spine plane block
  Other Names: 0.9% Sodium Chloride iv.
  Arms: placebo
Drug: Dexamethasone 4 Mg/mL Injectable Solution — biliteral administration of 20ml of 0,2% ropivacaine with 4mg Dexamethasone for the erector spine plane block
  Other Names: 0,2% ropivacaine with 4mg Dexamethasone iv
  Arms: Dexamethasone
Drug: Dexmedetomidine injection — biliteral administration of 20ml of 0,2% ropivacaine with 50ug Dexmedetomidine for the erector spine plane block
  Other Names: 0,2% ropivacaine with 50ug Dexmedetomidine
  Arms: Dexmedetomidine

SUMMARY:
Effect of perineurial dexamethasone and dexmedetomidine on erector spinal plane block duration for spine surgery.

DETAILED DESCRIPTION:
This study is proposed to explore the effect of perineurial Dexamethasone and Dexmedetomidine on erector spinal plane block duration for spine surgery.

After spine surgery, patients need good analgesia. Peripheral nerve blocks have provided a safe, effective method to control early postoperative pain when symptoms are most severe.

The safety of local anaesthesia is essential due to the much lower toxicity threshold of local anaesthetics. An effective adjuvant, such as Dexamethasone or Dexmedetomidine, could allow for a higher dilution of local anaesthetics while maintaining and enhancing their analgesic effect.

There is considerable research where intravenous and perineural dexamethasone and Dexmedetomidine use have been compared in adults. However, there is a massive lack of research regarding spine surgery and the Erector Spinae Plane Block.

In this study, investigators compare perineural Dexamethasone and Dexmedetomidine.

The investigator aims to find a dexamethasone or dexmedetomidine that covers the need for good pain relief and fast recovery postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing primary posterior lumbar decompression and stabilization with instrumentation involving multi-levels in the lumbar region,
* aged >18 years and <100 years
* ASA physical status 1, 2 or 3.

Exclusion Criteria:

* refuse to participate,
* history of opioid abuse,
* infection of the puncture site,
* aged <18 years and >100 years
* ASA 4 and 5

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
first need of opiate | 48 hours
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opioid consumption | 48 hours
  Total opiate consumption after surgery
Numerical Rating Scale [range 0:10] | Time Frame: 4 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | Time Frame: 8 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | Time Frame: 12 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | Time Frame: 16 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | Time Frame: 20 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
Numerical Rating Scale [range 0:10] | Time Frame: 24 hours after surgery
  NRS (Numerical Rating Scale; 0 - no pain; 10 - the worst pain ever)
NLR | 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
PLR | 48 hours after surgery
  Platelet-to-lymphocyte ratio

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Domagalska, PhD, Principal Investigator — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: No